CLINICAL TRIAL: NCT02841722
Title: Evaluation and Modeling of the G-CSF Effect on the Evolution of Neutrophils During Chemotherapy Based on Eribulin
Acronym: EMEG-E-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-A00123-46
Record Dates: First submitted 2016-04-21; First posted 2016-07-22 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biological samples (Other): Only one arm in this pilot study. All patient will have a follow up and treatment as per standard care for this pathology. Specifically for the study all patients will have 8 additional blood samples to be drawn during the first 2 cycles of treatment (1 cycles is 21 days).
  Interventions: Procedure: ERIBULIN + G-CSF (Granulocyte-Colony Stimulating Factor)

INTERVENTIONS:
Procedure: ERIBULIN + G-CSF (Granulocyte-Colony Stimulating Factor) — 8 additional blood samples

SUMMARY:
The anti-cancer cytotoxic chemotherapy is often the cause of neutropenia of grade IV or febrile neutropenia. Those neutropenia, in addition to being a comorbidity factor, result in dose reductions and/or temporary or permanent stop of chemotherapy, thus impacting clinical response. To avoid those episodes, or to shorten the duration and reduce the associated risk, administration of Granulocyte Colony Stimulating Factor (G-CSF) is recommended. Recombinant G-CSF reproduces the physiological effects of endogenous G-CSF by increasing the proliferation of granulocytes progenitors. Different forms of G-CSF are available: daily administration (such as filgrastim, lenograstim) and a single administration (pegfilgrastim).

Various international learned societies offer recommendations for primary care, secondary or curative neutropenia induced by chemotherapy based on G-CSF. However, guidance on the ideal time for the administration of growth factors and duration of administration are not very clear. If it seems clear that the treatment should not be initiated within the first 24 hours following administration of chemotherapy, summaries of the characteristics of different products do not provide evidence to optimize the administration day depending on the kinetics evolution of neutrophils. In addition, no information is given as to the choice of a formulation with respect to the other.

The pilot study the investigator propose aims to model the effect of exogenous G-CSF on the evolution of neutrophil function of time and explain the pharmacodynamic variability during the administration of chemotherapy based on eribulin. The description of the evolution of neutrophils when growth factors are administered give the opportunity to streamline administration regimens of these factors and to provide guidance on the circumstances in which they should or should not be given while weekly chemotherapy.

Expected benefits and foreseeable risks With the exception of surplus withdrawals during the first 2 cycles of treatment, this study will have no impact on the care of patients.

ELIGIBILITY:
Inclusion Criteria:

* Women
* over 18 years
* Patient with locally or metastatic advanced breast cancer histologically documented who received at least one chemotherapy regimen that includes an anthracycline and a taxane unless in patients who can not receive these treatments
* Patient to be treated with eribulin
* Patient that should preventively receive granulocyte growth factors at the first cycle (patient who already experienced febrile neutropenia, patient with a low neutrophil count at baseline, patient with a Performance Status altered or any other condition requiring administration of granulocyte colony stimulating factor as recommended by the oncologist)
* Neutrophils> 1500 / mm3; platelets> 100,000 / mm3
* Dated and signed Informed consent
* For patients of childbearing age, effective contraception during treatment and up to 3 months after stopping treatment

Exclusion Criteria:

* Patient with against-indication to treatment with eribulin such as hypersensitivity to the active substance or to any of the excipients, congenital long QT syndrome
* Patient already being treated with eribulin
* Patient with clinically detectable brain metastases
* Patient with against-indication to treatment with G-CSF such as hypersensitivity to the active substance or to any of the excipients
* Pregnant women or nursing
* Patient under guardianship or subject to major people protection regime
* Patient not affiliated with a social security scheme (beneficiary or beneficiary)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2015-12-03 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Variation of Neutrophils concentration in patient treated with G-CSF (Granulocyte-Colony Stimulating Factor) | Variation of Neutrophil concentration will be assess during the two first cycle of Eribulin treatment (1 cycle is 21 days, so total time frame is 42 days)
  variation of Neutrophil concentration will be assess by blood count formula performed during the 2 first cycle of Eribulin treatment: at the first and last day of G-CSF administration, at day 10 and day 15 of each cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle DESMOULINS, MD, Principal Investigator — Centre Georges François Leclerc
Locations (1):
- CGFL, Dijon, France

IPD SHARING:
Plan to Share IPD: No